CLINICAL TRIAL: NCT05310812
Title: Evaluation of Candidate Biomarkers to Predict Disease Severity and Acute Kidney Injury in Sepsis Patients in the Intensive Care Unit: Prospective Observational Study
Brief Title: Evaluation of Candidate Biomarkers to Predict Disease Severity and Acute Kidney Injury in Sepsis Patients
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mert CANBAZ, Principal Investigator M.D., Istanbul University
Other Study IDs: 2021/1907
Record Dates: First submitted 2022-02-27; First posted 2022-04-05 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Sepsis; Septic Shock; Acute Kidney Injury
Keywords: Sepsis; Acute Kidney Injury; Presepsin; Proenkefalin; Sindekan-1
MeSH Terms: conditions — Sepsis; Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group (Sepsis - no acute kindey injury): Septic patients diagnosed by sepsis criteria but no have an acute kidney injury. (According ot KDIGO classification - creatinin values).
  Blood plasma will be taken for biochemical evaluation.
  Interventions: Diagnostic Test: Biochemical evaluation.
- Study group (Sepsis induced acute kidney injury): Septic patients diagnosed by sepsis criteria, and have an acute kidney injury. (According ot KDIGO classification - creatinin values).
  Blood plasma will be taken for biochemical evaluation.
  Interventions: Diagnostic Test: Biochemical evaluation.

INTERVENTIONS:
Diagnostic Test: Biochemical evaluation. — Blood will be taken for biochemical evaluation-ELISA.
  Other Names: Presepsin; NGAL; Syndecan-1; Proencephalin

SUMMARY:
Investigators predict that the information that can be obtained in terms of renal functions before clinical development in sepsis patients can be valuable in terms of guiding treatment algorithms, planning renal replacement therapies and using drugs that are toxic to the kidneys.

DETAILED DESCRIPTION:
Despite the developments in Intensive Care Units (ICU), mortality and morbidity rates due to sepsis and septic shock are still high and it is seen as one of the major causes of death in ICU patients. Acute kidney injury (AKI) is a common disease worldwide and is seen in approximately 60% of intensive care hospitalizations. Diagnosis is generally made by the increase in serum creatinine level. Although it is a basic marker for AKI in current conditions, its levels can be misleading in clinical practice, especially in sepsis patients characterized by clinical conditions such as multiple organ failure. For these reasons, there is a need for new and applicable biomarkers that can be used in planning organ support treatments that can be applied to renal function in sepsis patients.

The utility of a new marker called presepsin in disease course, prognosis determination and sepsis-associated AKI clinic has been demonstrated. There are studies showing that neutrophil gelatinase-associated lipocalin (NGAL) is more valuable when compared to creatinine in patients with sepsis-associated AKI. Proenkephalin is a new biomarker studied, and it has been studied with NGAL in patients with cardiogenic shock, and it has been shown to have a place in the prediction of AKI in patients with cardiogenic shock. Significant elevation of syndecan-1 in acute kidney injury has been demonstrated in animal studies and clinical studies. In the literature, as far as investigators know, proenkephalin and syndecan-1 have not been studied in terms of AKI in sepsis patients.

In our study, investigators plan to investigate the role of biomarkers such as presepsin, syndecan-1, NGAL, and proenkephalin in predicting the risk of developing AKI in sepsis patients. The relevant markers will be studied from the blood sample taken from the patients diagnosed with sepsis at the time of diagnosis, and the results will be analyzed in terms of markers that may be more useful in predicting the development of AKI in patients. In addition, investigators aim to obtain clinical information by investigating whether these biomarkers have predictive properties on disease prognosis and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with sepsis and septic shock according to the "The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3)" guideline.
2. Signing of the Informed Consent Form by the patient or his legal representative.

Exclusion Criteria:

1. Patients under 18 years of age.
2. They are pregnant.
3. Malignant patients in the terminal period with no expected survival.
4. The Informed Consent Form is not signed by the patient or patient's relative.
5. Sepsis and septic shock patients admitted from another hospital under vasopressor or on mechanical ventilator.
6. Patients who develop brain damage and multi-organ failure after cardiopulmonary resuscitation.
7. Chronic renal failure patients receiving dialysis treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with sepsis and septic shock according to the "The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3)" guideline.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | 1st day in ICU
  KDIGO classification for acute kidney injury and biomarkers (ELISA test for Presepsin, Proencephalin, Syndecan-1 NGAL)
Mortality | 1st day in ICU
  Relationship between mortality rates and biomarkers (CRP, procalcitonin, white blood cell count, ELISA test for Presepsin, Proencephalin, Syndecan-1, NGAL.

SECONDARY OUTCOMES:
Disesase severity | 1st day in ICU
  Relationship between APACHE-SOFA scores and biomarkers (ELISA test for Presepsin, Proencephalin, Syndecan-1, NGAL)

CONTACTS AND LOCATIONS:
Overall Officials: Figen ESEN, Prof. Dr., Study Director — Istanbul University
Locations (1):
- Istanbul University, Istanbul Faculy of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No